CLINICAL TRIAL: NCT02244047
Title: Exploratory, Placebo-controlled Study on the Effects of Bifidobacterium Breve in Children With Celiac Disease
Brief Title: Cytokine Profile in Children With Celiac Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Martina Klemenak, medical doctor, resident at Pediatric department, University Medical Centre Maribor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEL-BIF
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacterium breve (Active Comparator): Bifidobacterium breve BR03 and B632 powder containing 10/9 CFU daily dosage in a period of 3 months
  Interventions: Drug: Bifidobacterium breve
- Placebo (Active Comparator): Placebo in the same powder packages as Bifidobacterium breve
  Interventions: Drug: Placebo (for Bifidobacterium breve)

INTERVENTIONS:
Drug: Bifidobacterium breve
  Arms: Bifidobacterium breve
Drug: Placebo (for Bifidobacterium breve)
  Arms: Placebo

SUMMARY:
Celiac disease (CD) is an immune-mediated systemic disease that is elicited by consumption of gluten and related prolamines in genetically susceptible individuals. Not only genetic but also environmental factors play an important role in CD pathogenesis. CD patients have imbalance in the gut microbiota, they have reduced number of Bididobacterium species in feces and biopsies.

Up till now, only effective treatment for CD is life long adherence to gluten free diet. If gluten free diet is not strict that leads over the years to complications of disease, such as autoimmune diseases, psychiatric diseases, osteoporosis etc. That may be caused by continuous recirculation of activated immune cells between the inflamed organ and the periphery. To avoid complications of disease in long term the investigators want to test specific probiotic bacteria from Bifidobacteria genus, that has has been in vitro studies recognized as anti-inflammatory.

Hypothesis

1. Children with celiac disease on gluten free diet have a higher level of pro-inflammatory cytokine (TNF-alpha) and anti-inflammatory cytokine (IL-10) in comparison with healthy controls.
2. 3 months after daily probiotic consumption TNF-alpha level decrease and IL-10 level increase.

In the investigators research will be selected 70 children, age from 2 to 18 years, divided in different groups:

1. Group: 25 children with celiac disease on GFD for at least 3 months and will receive probiotic for 3 months.
2. Group: 25 children with celiac disease on GFD for at least 3 months and will receive placebo for 3 months.
3. Group: 20 healthy children

ELIGIBILITY:
Inclusion Criteria:

* celiac disease on gluten free diet

Exclusion Criteria:

* acute or chronic diseases,
* permanent use of medication and
* ingestion of antibiotics at least one month prior to study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Serum TNF-alpha decrease after Bifidobacterium breve daily consumption in children with celiac disease | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Martina Klemenak, md, Principal Investigator — University Medical Centre Maribor

REFERENCES:
- [Derived] Klemenak M, Dolinsek J, Langerholc T, Di Gioia D, Micetic-Turk D. Administration of Bifidobacterium breve Decreases the Production of TNF-alpha in Children with Celiac Disease. Dig Dis Sci. 2015 Nov;60(11):3386-92. doi: 10.1007/s10620-015-3769-7. Epub 2015 Jul 2. PMID 26134988